CLINICAL TRIAL: NCT00485277
Title: A Phase I Trial of a Fixed Dose of MVA-BN-HER2 Following 1st- or 2nd-Line Chemotherapy for HER-2-Positive Metastatic Breast Cancer
Brief Title: A Safety and Immunology Study of a Modified Vaccinia Vaccine for HER-2(+) Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BNIT-BR-002
Record Dates: First submitted 2007-06-08; First posted 2007-06-12 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2010-09

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Vaccine; Metastatic; HER-2-positive; Phase I; HER-2 Positive Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: MVA-BN-HER2 — Experimental vaccine, subcutaneous injection q3weeks x 3

SUMMARY:
The current trial, BNIT-BR-002, will evaluate the safety and biological activity of a fixed dose of MVA-BN®-HER2, with and without Herceptin, following 1st- or 2nd-line chemotherapy in patients with Her-2-positive metastatic breast cancer.

The intent of vaccination is to induce anti-Her-2 immune responses, both antibody and T cell, that will then attack the Her-2 expressing tumors, and may induce tumor regression or slow progression of disease.

DETAILED DESCRIPTION:
MVA-BN®-HER2 is a candidate breast cancer immunotherapy product comprised of a highly attenuated non-replicating vaccinia virus, MVA-BN®, engineered to encode a modified form of the Her-2 protein.

MVA-BN® is a well-characterized, clonal strain of modified vaccinia virus Ankara (MVA) being developed as a smallpox vaccine, suitable for use in high-risk (e.g., immunocompromised) individuals. MVA-BN®-derived vectors encoding heterologous antigens are being developed for use as vaccines for infectious diseases such as HIV, and for the treatment of cancer. A large database exists from safety evaluations in animals and in humans for MVA-BN®, and MVA-BN®-derived vectors.

Her-2 is overexpressed in 20-30% of human breast cancers. It is an oncogene/growth factor receptor critical for malignant phenotype of Her-2 expressing tumors. It is an immunogenic target, and immune responses to this protein have been shown to mediate potent anti-tumor activity in multiple animal models. Means to stimulate anti-Her-2 reactivity are now being studied clinically. Sponsor, collaborators, and others have used both Protein and DNA vaccine forms of Her-2, and a safety database is developed and no significant adverse events have resulted from Her-2 directed vaccination.

MVA-BN®-HER2 encodes a modified form of the Her-2 protein, hereinafter referred to as HER2. HER2 contains the extracellular domain of Her-2 but lacks the intracellular, cell signaling domain. In addition, HER2 includes two universal T-cell epitopes from tetanus toxin to facilitate the stimulation of an immune response to Her-2, a self-protein.

The current trial, BNIT-BR-002, will evaluate the safety and biological activity of a fixed dose of MVA-BN®-HER2, with and without Herceptin, following 1st- or 2nd-line chemotherapy in patients with metastatic breast cancers which overexpress Her-2.

Patients will receive 3 subcutaneous vaccinations at 3 week intervals and have tumor followed by CT/MRI imaging and blood drawn for immune function analysis.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Women, ≥ 18 years of age
* Histologically documented, HER-2 (+) breast cancer with metastatic disease.
* Evaluable or measurable disease. PATIENTS MAY BE NED. Patients must be assessed as having stable disease or better at the end of 1st- or 2nd-line chemotherapy. In addition, patients must have a tumor assessment within 28 days of the first planned dose of MVA-BN®-HER2, and have a response status of SD or better.
* Prior chemotherapy for metastatic breast cancer
* Completed 1st- or 2nd-line chemo for mBrCA at least 3 weeks (from the date of the last dose) prior to the first dose of MVA-BN®-HER2
* ECOG Performance Score of 0, 1, or 2
* Life expectancy ≥ 6 months
* Left ventricular ejection fraction (LVEF) by ECHO or MUGA ≥ LLN
* Women of childbearing potential must have a negative serum or urine pregnancy test, and must agree to use a medically acceptable barrier and/or chemical method of contraception throughout the study treatment period and for 28 days after the last dose of MVA-BN®-HER2
* No significant cardiac, bone marrow dysfunction, or coagulopathy. No significant hepatic or renal dysfunction.
* A negative virology screen for HIV, hepatitis B surface antigen, hepatitis C, and HTLV-1

Exclusion Criteria:

Patients may not have:

* Known history of metastasis to the central nervous system
* Congestive heart failure (NYHA Class III or IV), unstable angina, or cardiovascular disease such as stroke or myocardial infarction (current or within the past 6 months)
* History of prior malignancies other than breast cancer within the past 5 years, excluding basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Known allergy to eggs, egg products, or aminoglycoside antibiotics, e.g., gentamicin or tobramycin
* Chronic administration (5 or more consecutive days) of systemic corticosteroids within 14 days of the first planned dose of MVA-BN®-HER2.
* History of or active autoimmune disease. Persons with vitiligo or thyroid disease taking thyroid replacement hormones are not excluded.
* Prior solid organ or hematopoietic allogenic transplant(s)
* Prior use of hematopoietic growth factors (e.g., GM-CSF) within 28 days of the first planned dose of MVA-BN®-HER2
* Receipt of an investigational agent within 28 days of the first planned dose of MVA-BN®-HER2
* Prior "vaccine" therapy for breast cancer at any time
* Vaccination: Vaccinations with a live (attenuated) vaccine within 28 days of the first or last dose of study drug; or vaccinations with a killed (inactivated) vaccine within 14 days of the first or last dose of study drug.
* A maximum cumulative dose of prior doxorubicin > 360 mg/m2 or epirubicin > 720 mg/m2
* Radiation therapy within 28 days of the first planned dose of MVA-BN®-HER2 or plans for radiation therapy after enrollment.
* Pregnant, lactating, or nursing
* Any condition which, in the opinion of the investigator, would prevent full participation in this trial or the long-term follow-up study, or would interfere with the evaluation of the trial endpoints

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 2years, 3 months

SECONDARY OUTCOMES:
Immune response | 2 yrs 3 mo

CONTACTS AND LOCATIONS:
Overall Officials: Olga Bandman, Study Director — Bavarian Nordic
Locations (2):
- United States (2):
  - Alta Bates Herrick Hospital Comprehensive Cancer Center, Berkeley, California
  - Stanford Cancer Center, Stanford, California